CLINICAL TRIAL: NCT00491556
Title: Preservation and Expansion of T-cell Subsets Following HAART De-intensification to Atazanavir/Ritonavir (ATV/r) in Adolescents With CD4 + T Cells > 350 Cells/mm3 Initiating HAART
Brief Title: Preservation and Expansion of T-cell Subsets Following HAART De-intensification to Atazanavir/Ritonavir (ATV/r)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN 061
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2016-05

CONDITIONS: HIV Infections
Keywords: Atazanavir/Ritonavir (ATV/r); highly-active antiretroviral therapy (HAART); Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm (Experimental): Subjects in the experimental group will begin HAART consisting of TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r or other recommended NRTI backbone with ATV/r upon entry or to begin treatment under current DHHS guidelines. Subjects in the experimental group who achieve virologic control by week 24 and maintain good control through 48 weeks will then de-intensify to ATV/r alone and will be followed for an additional two years.
  Interventions: Procedure: Early Initiation of Highly Active Anti-Retroviral Therapy
- Standard Care Arm (Other): Subjects randomized to the standard care arm will begin HAART with TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r, or other recommended ATV/r based HAART regimen according to current DHHS standard of care and will be followed for a total of three years. Under these guidelines and under current clinical standards, subjects on the standard care arm will begin therapy when the CD4+ T cell count drops below 350 cells/mm3 or other clinical criteria necessitating treatment as determined by the site clinician occur.
  Interventions: Procedure: Standard Care

INTERVENTIONS:
Procedure: Early Initiation of Highly Active Anti-Retroviral Therapy — Treatment: TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r or other recommended NRTI backbone with ATV/r. Duration: Subjects in the experimental group who achieve virologic control by week 24 and maintain good control through 48 weeks will then de-intensify to ATV/r alone and will be followed for an additional two years.
  Arms: Experimental Arm
Procedure: Standard Care — Progression: Subjects on the standard care arm will begin therapy when the CD4+ T cell count drops below 350 cells/mm3 or other clinical criteria necessitating treatment as determined by the site clinician occur. Treatment: HAART with TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r, or other recommended ATV/r based HAART regimen according to current DHHS standard of care. Duration: three years.
  Arms: Standard Care Arm

SUMMARY:
This study proposes to evaluate a pre-DHHS guideline of HAART initiation and then de-intensification management strategy in adolescents with mild immunosuppression and compare changes in CD4% from baseline to week 48 and then during de-intensification.

DETAILED DESCRIPTION:
This is a randomized, proof of concept study of youth 18- 24 years of age with confirmed HIV after age 9 with CD4+ T cells above 350 cells/mm3 who are randomized 3:1 to begin HAART consisting of TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r, or other recommended NRTI backbone with ATV/r upon entry or to begin treatment under current DHHS guidelines. Subjects in the experimental group who achieve virologic control by week 24 and maintain good control through 48 weeks will then de-intensify to ATV/r alone and will be followed for two years. Subjects randomized to the standard care arm will begin HAART with TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r, or other recommended ATV/r based HAART regimen according to current DHHS standard of care.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 yrs and 0 days to 24 yrs and 364 days;
2. CD4+ T cells > 350/mm3 and HIV RNA ≥ 1,000 copies/ml as determined by two consecutive measures within 6 months of entry with the second measure being collected at pre-entry;
3. Infected after age 9. HIV-1 infection should be documented by any licensed ELISA test kit and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA at any time prior to entry; Note: Subjects who are in acute seroconversion as evidenced by being ELISA negative (antibody negative) and DNA PCR or HIV-1 RNA positive or who are ELISA positive but Western Blot indeterminate are not eligible.
4. Subjects must be naïve to ARV medications except for women who have received HAART for prevention of maternal to child transmission (MTCT) that meet the following criteria: HAART (defined as three medications from two classes) given for no more than six months for prevention of MTCT, Evidence of viral suppression on the HAART regimen defined as a plasma RNA level below the level of detection for the assay used by the site either during the third trimester or around the time of delivery, A minimum of six months since HAART exposure for prevention of MTCT, and Exposure to HAART for a single pregnancy only; Note: Prior treatment with Trizivir for prevention of MCTC is also permitted as long as viral suppression is documented at the time of delivery or in the last trimester, whichever is most recent.
5. HIV genotype without major resistance mutations to ATV/r. The following genotypic mutations exclude subjects from participation in ATN 061: Major ATV mutations I50L; I84V; N88D/S, Major PI mutations including: D30N; V32I; L33I/F/V; M46I/L; I47V/A; G48V; I50V/L; I54V/L/A/M/T/S; L76V; V82A/F/T/S/L; L90M, Any major PI mutation as defined by the most current IAS-USA Drug Resistance Mutations Figures that would adversely affect a subject's future PI choices, Major RT mutations: Q151M and 69 insertion complex; Decisions regarding the selection of an NRTI backbone for subjects with NRTI resistance mutations other than those described above will be made by the site PI in consultation with the protocol chair or his designee. Whenever possible and not otherwise contraindicated, NRTI choices should be congruent with the protocol-specified preferred regimens. The site PI must provide a copy of the genotype analysis along with their proposed regimen for review; Note: Subjects who cannot go onto either FTC/TDF or AZT/3TC must have the regimen approved by the protocol team following pre-entry screening and prior to study entry. Note: All HIV-1 genotype profiles with ANY resistance mutations must be evaluated by a physician specializing in the care of HIV-infected patients prior to final determination of subject eligibility. Polymorphism mutations should NOT be reported since their clinical significance is unknown. All other (major and minor) mutations should be appropriately categorized and reported as indicated by the case report form. In circumstances where there are numerous such mutations or other concerns present, consultation with the protocol team by the evaluating physician via the ATN QNS is highly encouraged.
6. Calculated creatinine clearance ≥60 mL/min as estimated by the Cockcroft-Gault equation: For men, (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72) = CrCl (mL/min)*;*For women, multiply the result by 0.85 = CrCl (mL/min);
7. For females with child-bearing potential, agreement to use one effective birth control method and willing to postpone pregnancy for the duration of the study (See Section 9.3 - criteria for class C drugs should be followed); and
8. Able to provide written informed consent/assent.

Exclusion Criteria

1. Pregnancy;
2. On systemic immunosuppressive therapy or immune modulating therapy (short courses (<14 days) of prednisone for reactive airway disease [RAD] are permitted but not within 30 days prior to study entry);
3. Any history of an AIDS-defining illness (note: a history of a CD4 + T cell count below 200 cells/mm3 is not an exclusion criterion as long as all other inclusion/exclusion criteria are met);
4. Currently breast feeding;
5. Current treatment for active serious systemic bacterial infections;
6. Active hepatitis B infection as defined by Hepatitis B Ag positive;
7. Treatment with immune modulators including IL-2, intravenous gammaglobulin, and therapeutic or other experimental vaccines including HIV-1 vaccine given for primary prevention at any time;
8. History of cardiac conduction abnormalities including one or more of the following: Symptomatic heart block, Third-degree heart block, even if asymptomatic, Pre-excitation syndromes, Heart Rate <40 bpm, Ventricular pause length >3 seconds, QTc > 500 msec, and Cardiomyopathy;
9. Disallowed Medications (see Section 5.3.2);
10. Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with adherence to the study;
11. History of chronic renal insufficiency or Grade 3 or greater serum creatinine; and
12. Any confirmed grade 3 or greater laboratory value at pre-entry (with the exception of grade 3 or greater lipids or platelets).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2007-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret J Rudy, M.D., Study Chair — Children's Hospital of Philadelphia; John Sleasman, M.D., Study Chair — University of South Florida, Dept of Pediatrics
Locations (23):
- United States (22):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - University of Southern California - IMPAACT Site, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital of Denver - IMPAACT Site, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University - IMPAACT Site, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of Southern Florida College of Medicine, Tampa, Florida
  - Stoger Hospital of Cook County, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University - IMPAACT Site, Baltimore, Maryland
  - Children's Hospital of Michigan - IMPAACT Site, Detroit, Michigan
  - UMDNJ - IMPAACT Site, Newark, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Pediatric Infectious Diseases - IMPAACT Site, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital (Memphis) - IMPAACT Site, Memphis, Tennessee
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Borkar SA, Yin L, Venturi GM, Shen J, Chang KF, Fischer BM, Nepal U, Raplee ID, Sleasman JW, Goodenow MM. Youth Who Control HIV on Antiretroviral Therapy Display Unique Plasma Biomarkers and Cellular Transcriptome Profiles Including DNA Repair and RNA Processing. Cells. 2025 Feb 15;14(4):285. doi: 10.3390/cells14040285. PMID 39996757
- See also: Description of Adolescent Trials Networks (ATN) and contact information — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research was conducted at 23 clinical sites. Accrual was open between August 2007 and June 2010.
Groups:
- Experimental-Early Initiation of HAART (EXP): Began HAART consisting of TDF/FTC/ATV/r (preferred regimen), AZT/3TC/ATV/r, or other recommended NRTI HAART backbone with ATV/r upon entry to study. Subjects who achieved virologic control by week 24 (viral load (VL) < 100 copies/ml) and maintained good control through 48 weeks then entered deintensification (de-int) to ATV/r alone and were followed for two years.
- Standard Care (STAND): Began HAART with ATV/r under the current DHHS guidelines (CD4+ T cells below 350 cells/mm3 or for other clinical concerns as outlined in the recommendations and as determined by the site clinician).
Period: Entry-Week (WK) 48: EXP/Standard Care
Arm/Group | Experimental-Early Initiation of HAART (EXP) | Standard Care (STAND)
Started | 75 | 27
Wk 24 VL Suppressed (EXP)/WK 24 (STAND) | 53 | 27
Completed | 49 | 27
Not Completed | 26 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Moved Out of Area | 2 | 0
Not completed — Failure to Suppress VL at Week 24 | 11 | 0
Not completed — VL Failure at Week 24 | 2 | 0
Not completed — Adherence Issues | 2 | 0
Not completed — Toxicity | 3 | 0
Not completed — Other | 3 | 0
Period: Wk 48-152: EXP (On De-Int)/Standard Care
Arm/Group | Experimental-Early Initiation of HAART (EXP) | Standard Care (STAND)
Started | 49 | 27
Completed | 25 | 22
Not Completed | 24 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Pregnancy | 2 | 0
Not completed — Moved Out of Area | 2 | 1
Not completed — VL Failure After Week 48 | 5 | 0
Not completed — CD4 Failure | 2 | 0
Not completed — Adherence Issues | 5 | 0
Not completed — Toxicity | 2 | 0
Not completed — End of Funding | 2 | 0
Not completed — Other | 2 | 0
Not completed — Incarceration | 0 | 1
Not completed — Death of Participant | 0 | 1

BASELINE CHARACTERISTICS:
Population: 75 subjects were randomized to the experimental arm, however 2 subjects withdrew from the study at the pre-entry visit. Therefore, only 73 experimental arm subjects were available for the baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Standard Care Arm | Total
Number analyzed (Participants) | 73 | 27 | 100
Age, Customized [Number; unit: participants]
  18-20 years | 31 | 10 | 41
  21-24 years | 42 | 17 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 64 | 23 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 6 | 0 | 6
  Black non-Hispanic | 47 | 23 | 70
  Hispanic | 17 | 2 | 19
  Asian | 2 | 1 | 3
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 72 | 27 | 99
  Puerto Rico | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference in CD4+ T Cell Percentage Between Week 0 and Week 48
Time Frame: Week 0 and Week 48
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized to the experimental arm.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T cells
Groups:
- Experimental-Early Initiation of HAART (EXP): Subjects in the experimental group will begin HAART consisting of TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r or other recommended NRTI backbone with ATV/r upon entry or to begin treatment under current DHHS guidelines. Subjects in the experimental group who achieve virologic control by week 24 and maintain good control through 48 weeks will then de-intensify to ATV/r alone and will be followed for an additional two years.
  Early Initiation of Highly Active Anti-Retroviral Therapy: Treatment: TDF/FTC/ATV/r (preferred), AZT/3TC/ATV/r or other recommended NRTI backbone with ATV/r. Duration: Subjects in the experimental group who achieve virologic control by week 24 and maintain good control through 48 weeks will then de-intensify to ATV/r alone and will be followed for an additional two years.
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 25
percentage of CD4+ T cells | -10.08 (5.13)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -10.08, 95% CI 2-sided [-12.20 to -7.97], Standard Deviation 5.13 — Difference was calculated as Baseline minus Week 48

2. Primary Outcome: Difference in CD4+ T Cell Percentage Between Week 48 and Week 152
Time Frame: 152 Weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 25
percentage of CD4+ T cells | -1.81 (5.00)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0834, t-test, 2 sided; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-3.87 to 0.26], Standard Deviation 5.00 — Difference was calculated as Week 48 minus Week 152

3. Secondary Outcome: Difference in CD4+ T Cell Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: CD4+ T cells/cubic millimeter
Arm/Group | Experimental Arm
Number analyzed (Participants) | 25
CD4+ T cells/cubic millimeter | -317.36 (176.07)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -317.36, 95% CI 2-sided [-390.04 to -244.68], Standard Deviation 176.07 — Difference was calculated as Baseline minus Week 48

4. Secondary Outcome: Difference in CD4+ T Cell Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: CD4+ T cells/cubic millimeter
Arm/Group | Experimental Arm
Number analyzed (Participants) | 25
CD4+ T cells/cubic millimeter | -24.20 (242.38)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.6222, t-test, 2 sided; Mean Difference (Final Values) = -24.20, 95% CI 2-sided [-124.25 to 75.85], Standard Deviation 242.38 — Difference was calculated as Week 48 minus Week 152

5. Secondary Outcome: Difference in CD4+ Naïve T Cell Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm.Two subjects did not have enough blood samples to measure CD4+ Naïve T-Cell count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD4+ naïve t-cells/cubic millimeter
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
CD4+ naïve t-cells/cubic millimeter | -58.79 (152.57)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.0781, t-test, 2 sided; Mean Difference (Final Values) = -58.79, 95% CI 2-sided [-124.77 to 7.18], Standard Deviation 152.57

6. Secondary Outcome: Difference in CD4+ Naïve T Cell Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: CD4+ naïve t-cells/cubic millimeter
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
CD4+ naïve t-cells/cubic millimeter | -103.53 (176.61)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0102, t-test, 2 sided; Mean Difference (Final Values) = -103.53, 95% CI 2-sided [-179.90 to -27.16], Standard Deviation 176.61

7. Secondary Outcome: Difference in CD4+ Termed Central Memory (TCM) Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm.Two subjects did not have enough blood samples to measure CD4+ Termed Central Memory (TCM) count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD4+ TCM cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD4+ TCM cells/cubic millimeter | -17.13 (56.72)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.1616, t-test, 2 sided; Mean Difference (Final Values) = -17.13, 95% CI 2-sided [-41.66 to 7.40], Standard Deviation 56.72 — Difference was calculated as Baseline minus Week 48

8. Secondary Outcome: Difference in CD4+ TCM Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm.Two subjects did not have enough blood samples to measure CD4+ TCM count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD4+ TCM cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD4+ TCM cells/cubic millimeter | -43.08 (75.17)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0117, t-test, 2 sided; Mean Difference (Final Values) = -43.08, 95% CI 2-sided [-75.59 to -10.58], Standard Deviation 75.17 — Difference was calculated as Week 48 minus Week 152

9. Secondary Outcome: Difference in CD4+ Effector Memory (TEM)Ro Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD4+ Effector Memory (TEM)Ro count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD4+ TemRo cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD4+ TemRo cells/cubic millimeter | -76.92 (56.31)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -76.92, 95% CI 2-sided [-101.27 to -52.57], Standard Deviation 56.31 — Difference was calculated as Baseline minus Week 48

10. Secondary Outcome: Difference in CD4+ TEMRo Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD4+ TEMRo count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD4+ TemRo cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD4+ TemRo cells/cubic millimeter | 16.87 (68.75)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.2519, t-test, 2 sided; Mean Difference (Final Values) = 16.87, 95% CI 2-sided [-12.86 to 46.60], Standard Deviation 68.75 — Difference was calculated as Week 48 minus Week 152

11. Secondary Outcome: Difference in CD4+ TEMRa Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD4+ TEMRa count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD4+ TEMRa cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD4+ TEMRa cells/cubic millimeter | -126.79 (105.61)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -126.79, 95% CI 2-sided [-172.46 to -81.12], Standard Deviation 105.61 — Difference was calculated as Baseline minus Week 48

12. Secondary Outcome: Difference in CD4+ TEMRa Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: CD4+ TEMRa cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD4+ TEMRa cells/cubic millimeter | 87.64 (97.71)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided; Mean Difference (Final Values) = 87.64, 95% CI 2-sided [45.39 to 129.90], Standard Deviation 97.71 — Difference was calculated as Week 48 minus Week 152

13. Secondary Outcome: Difference in CD8+ Naïve T-Cell Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8+ Naïve T-Cell count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD8+ naïve t-cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ naïve t-cells/cubic millimeter | 40.46 (213.77)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.3739, t-test, 2 sided; Mean Difference (Final Values) = 40.46, 95% CI 2-sided [-51.98 to 132.90], Standard Deviation 213.77 — Difference was calculated as Baseline minus Week 48

14. Secondary Outcome: Difference in CD8+ Naïve T-Cell Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: CD8+ naïve T cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ naïve T cells/cubic millimeter | -91.86 (166.40)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0147, t-test, 2 sided; Mean Difference (Final Values) = -91.86, 95% CI 2-sided [-163.82 to -19.90], Standard Deviation 166.40 — Difference was calculated as Week 48 minus Week 152

15. Secondary Outcome: Difference in CD8+ TCM Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8+ TCM count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD8+ TCM cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ TCM cells/cubic millimeter | 79.81 (76.07)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 79.81, 95% CI 2-sided [46.92 to 112.71], Standard Deviation 76.07 — Difference was calculated as Baseline minus Week 48

16. Secondary Outcome: Difference in CD8+ TCM Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: CD8+ TCM cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ TCM cells/cubic millimeter | -20.40 (58.18)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.1067, t-test, 2 sided; Mean Difference (Final Values) = -20.40, 95% CI 2-sided [-45.56 to 4.76], Standard Deviation 58.18 — Difference was calculated as Week 48 minus Week 152

17. Secondary Outcome: Difference in CD8+ TEMRo Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8+ TEMRo count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD8+ TEMRo cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ TEMRo cells/cubic millimeter | 90.82 (107.80)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.0005, t-test, 2 sided; Mean Difference (Final Values) = 90.82, 95% CI 2-sided [44.20 to 137.43], Standard Deviation 107.80 — Difference was calculated as Baseline minus Week 48

18. Secondary Outcome: Difference in CD8+ TEMRo Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: CD8+ TEMRo cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ TEMRo cells/cubic millimeter | 33.49 (64.41)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0207, t-test, 2 sided; Mean Difference (Final Values) = 33.49, 95% CI 2-sided [5.64 to 61.34], Standard Deviation 64.41 — Difference was calculated as Week 48 minus Week 152

19. Secondary Outcome: Difference in CD8+ TEMRa Count Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8+ TEMRa count, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: CD8+ TEMRa cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ TEMRa cells/cubic millimeter | -39.37 (145.62)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.2082, t-test, 2 sided; Mean Difference (Final Values) = -39.37, 95% CI 2-sided [-102.34 to 23.60], Standard Deviation 145.62 — Difference was calculated as Baseline minus Week 48

20. Secondary Outcome: Difference in CD8+ TEMRa Count Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: CD8+ TEMRa cells/cubic millimeter
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
CD8+ TEMRa cells/cubic millimeter | 48.27 (139.33)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0067, t-test, 2 sided; Mean Difference (Final Values) = 86.98, 95% CI 2-sided [26.73 to 147.23], Standard Deviation 139.33 — Difference was calculated as Week 48 minus Week 152

21. Secondary Outcome: Difference in CD8 Naïve CD28 Cell Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 Naïve CD28 Cell percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 naïve CD28 cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 naïve CD28 cells | -18.07 (13.20)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -18.07, 95% CI 2-sided [-23.78 to -12.36], Standard Deviation 13.20 — Difference was calculated as Baseline minus Week 48

22. Secondary Outcome: Difference in CD8 Naïve CD28 Cell Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage of CD8 Naïve CD28 Cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 Naïve CD28 Cells | 1.66 (14.20)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.5815, t-test, 2 sided; Mean Difference (Final Values) = 1.66, 95% CI 2-sided [-4.48 to 7.80], Standard Deviation 14.20 — Difference was calculated as Week 48 minus Week 152

23. Secondary Outcome: Difference in CD8 Naïve CD38 Cell Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 Naïve CD38 Cell percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 naïve CD38 cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 naïve CD38 cells | 11.24 (7.82)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 11.24, 95% CI 2-sided [7.85 to 14.62], Standard Deviation 7.82 — Difference was calculated as Baseline minus Week 48

24. Secondary Outcome: Difference in CD8 Naïve CD38 Cell Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percentage of CD8 naïve CD38 cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 naïve CD38 cells | -2.87 (6.93)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0594, t-test, 2 sided; Mean Difference (Final Values) = -2.87, 95% CI 2-sided [-5.87 to 0.12], Standard Deviation 6.93 — Difference was calculated as Week 48 minus Week 152

25. Secondary Outcome: Difference in CD8 Naïve CD57 Cell Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 Naïve CD57 Cell percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 naïve CD57 cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 naïve CD57 cells | 12.58 (10.24)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 12.58, 95% CI 2-sided [8.15 to 17.01], Standard Deviation 10.24 — Difference was calculated as Baseline minus Week 48

26. Secondary Outcome: Difference in CD8 Naïve CD57 Cell Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: percentage of CD8 naïve CD57 cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 naïve CD57 cells | 3.93 (10.95)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0995, t-test, 2 sided; Mean Difference (Final Values) = 3.93, 95% CI 2-sided [-0.81 to 8.66], Standard Deviation 10.95 — Difference was calculated as Week 48 minus Week 152

27. Secondary Outcome: Difference in CD8 Naïve T-Cell Percentage Expressing Human Leukocyte Antigen-D Related (HLA-DR) Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 Naïve T-Cell percentage Expressing Human Leukocyte Antigen-D related (HLA-DR), therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 naïve HLA-DR T-cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 naïve HLA-DR T-cells | 1.95 (2.07)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided; Mean Difference (Final Values) = 1.95, 95% CI 2-sided [1.05 to 2.84], Standard Deviation 2.07 — Difference was calculated as Baseline minus Week 48

28. Secondary Outcome: Difference in CD8 Naïve T-Cell Percentage Expressing HLA-DR Between Week 48 and Week 152
Time Frame: 152 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 Naïve T-Cell percentage Expressing HLA-D, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 naïve HLA-DR T cells
Arm/Group | Experimental-Early Initiation of HAART (EXP)
Number analyzed (Participants) | 23
percentage of CD8 naïve HLA-DR T cells | 0.03 (1.49)
Statistical Analysis 1: Comparison: Experimental-Early Initiation of HAART (EXP); Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.9150, t-test, 2 sided; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.61 to 0.68], Standard Deviation 1.49 — Difference was calculated as Week 48 minus Week 152

29. Secondary Outcome: Difference in CD8 TCM CD28 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TCM CD28 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM CD28 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM CD28 cells | -23.52 (13.79)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -23.52, 95% CI 2-sided [-29.48 to -17.55], Standard Deviation 13.79 — Difference was calculated as Baseline minus Week 48

30. Secondary Outcome: Difference in CD8 TCM CD28 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM CD28 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM CD28 cells | 1.95 (16.96)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.5864, t-test, 2 sided; Mean Difference (Final Values) = 1.95, 95% CI 2-sided [-5.38 to 9.28], Standard Deviation 16.96 — Difference was calculated as Week 48 minus Week 152

31. Secondary Outcome: Difference in CD8 TCM CD38 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TCM CD38 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM CD38 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM CD38 cells | 21.98 (8.48)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 21.98, 95% CI 2-sided [18.31 to 25.65], Standard Deviation 8.48 — Difference was calculated as Baseline minus Week 48

32. Secondary Outcome: Difference in CD8 TCM CD38 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM CD38 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM CD38 cells | -2.20 (7.25)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.1592, t-test, 2 sided; Mean Difference (Final Values) = -2.20, 95% CI 2-sided [-5.34 to 0.93], Standard Deviation 7.25 — Difference was calculated as Week 48 minus Week 152

33. Secondary Outcome: Difference in CD8 TCM CD57 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TCM CD57 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM CD57 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM CD57 cells | 4.97 (11.04)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.0420, t-test, 2 sided; Mean Difference (Final Values) = 4.97, 95% CI 2-sided [0.20 to 9.74], Standard Deviation 11.04 — Difference was calculated as Baseline minus Week 48

34. Secondary Outcome: Difference in CD8 TCM CD57 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM CD57 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM CD57 cells | -2.20 (12.39)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.4029, t-test, 2 sided; Mean Difference (Final Values) = -2.20, 95% CI 2-sided [-7.56 to 3.16], Standard Deviation 12.39 — Difference was calculated as Week 48 minus Week 152

35. Secondary Outcome: Difference in CD8 TCM HLA-DR Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TCM HLA-DR percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM HLA-DR T cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM HLA-DR T cells | 14.60 (6.03)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 14.60, 95% CI 2-sided [11.99 to 17.21], Standard Deviation 6.03 — Difference was calculated as Baseline minus Week 48

36. Secondary Outcome: Difference in CD8 TCM HLA-DR Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: percentage of CD8 TCM HLA-DR T cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TCM HLA-DR T cells | -3.14 (6.20)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0239, t-test, 2 sided; Mean Difference (Final Values) = -3.14, 95% CI 2-sided [-5.81 to -0.46], Standard Deviation 6.20 — Difference was calculated as Week 48 minus Week 152

37. Secondary Outcome: Difference in CD8 TEMRo CD28 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRo CD28 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRo CD28 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRo CD28 cells | -19.35 (10.26)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -19.35, 95% CI 2-sided [-23.79 to -14.91], Standard Deviation 10.26 — Difference was calculated as Baseline minus Week 48

38. Secondary Outcome: Difference in CD8 TEMRo CD28 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRo CD28 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRo CD28 cells | -3.45 (13.60)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.2363, t-test, 2 sided; Mean Difference (Final Values) = -3.45, 95% CI 2-sided [-9.33 to 2.43], Standard Deviation 13.60 — Difference was calculated as Week 48 minus Week 152

39. Secondary Outcome: Difference in CD8 TEMRo CD38 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRo CD38 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRo CD38 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRo CD38 cells | 19.69 (8.70)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 19.69, 95% CI 2-sided [15.93 to 23.45], Standard Deviation 8.70 — Difference was calculated as Baseline minus Week 48

40. Secondary Outcome: Difference in CD8 TEMRo CD38 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRo CD38 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRo CD38 cells | -2.03 (5.55)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0929, t-test, 2 sided; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-4.43 to 0.37], Standard Error of Mean 5.55 — Difference was calculated as Week 48 minus Week 152

41. Secondary Outcome: Difference in CD8 TEMRo CD57 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRo CD57 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRo CD57 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRo CD57 cells | -2.53 (8.94)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.1886, t-test, 2 sided; Mean Difference (Final Values) = -2.53, 95% CI 2-sided [-6.40 to 1.34], Standard Deviation 8.94 — Difference was calculated as Baseline minus Week 48

42. Secondary Outcome: Difference in CD8 TEMRo CD57 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRo CD57 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRo CD57 cells | 1.87 (8.13)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.2831, t-test, 2 sided; Mean Difference (Final Values) = 1.87, 95% CI 2-sided [-1.65 to 5.38], Standard Deviation 8.13 — Difference was calculated as Week 48 minus Week 152

43. Secondary Outcome: Difference in CD8 TEMRO HLADR Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRO HLADR percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRO HLADR
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRO HLADR | 11.52 (5.59)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 11.52, 95% CI 2-sided [9.10 to 13.94], Standard Deviation 5.59 — Difference was calculated as Baseline minus Week 48

44. Secondary Outcome: Difference in CD8 TEMRo HLA-DR Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRo HLA-DR percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRo HLA-DR cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRo HLA-DR cells | -3.21 (5.88)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0157, t-test, 2 sided; Mean Difference (Final Values) = -3.21, 95% CI 2-sided [-5.75 to -0.67], Standard Deviation 5.88 — Difference was calculated as Week 48 minus Week 152

45. Secondary Outcome: Difference in CD8 TEMRa CD28 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm.Three subjects did not have enough blood samples to measure CD8 TEMRa CD28 percentage, therefore the number of participants analyzed was reduced from 25 to 22 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TemRA CD28 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 22
percentage of CD8 TemRA CD28 cells | -22.65 (12.93)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -22.65, 95% CI 2-sided [-28.24 to -17.06], Standard Deviation 12.93 — Difference was calculated as Baseline minus Week 48

46. Secondary Outcome: Difference in CD8 TEMRa CD28 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm.Two subjects did not have enough blood samples to measure CD8 TEMRa CD28 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRa CD28 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRa CD28 cells | 4.23 (15.37)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.1999, t-test, 2 sided; Mean Difference (Final Values) = 4.23, 95% CI 2-sided [-2.41 to 10.88], Standard Deviation 15.37 — Difference was calculated as Week 48 minus Week 152

47. Secondary Outcome: Difference in CD8 TEMRa CD38 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRa CD38 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRa CD38 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRa CD38 cells | 12.47 (6.81)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 12.47, 95% CI 2-sided [9.52 to 15.41], Standard Deviation 6.81 — Difference was calculated as Baseline minus Week 48

48. Secondary Outcome: Difference in CD8 TEMRa CD38 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRa CD38 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRa CD38 cells | -1.95 (5.12)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0808, t-test, 2 sided; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-4.17 to 0.26], Standard Deviation 5.12 — Difference was calculated as Week 48 minus Week 152

49. Secondary Outcome: Difference in CD8 TEMRa CD57 Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRa CD57 percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRa CD57 cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRa CD57 cells | 11.70 (13.83)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p = 0.0005, t-test, 2 sided; Mean Difference (Final Values) = 11.70, 95% CI 2-sided [5.72 to 17.69], Standard Deviation 13.83 — Difference was calculated as Baseline minus Week 48

50. Secondary Outcome: Difference in CD8 TEMRa CD57 Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRa CD57cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRa CD57cells | -0.30 (14.12)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.9198, t-test, 2 sided; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-6.41 to 5.81], Standard Deviation 14.12 — Difference was calculated as Week 48 minus Week 152

51. Secondary Outcome: Difference in CD8 TEMRa HLA-DR Percentage Between Week 0 and Week 48
Time Frame: 48 weeks
Population: Subjects who maintained viral load suppression from Week 24 to Week 152 among those randomized in to the experimental arm. Two subjects did not have enough blood samples to measure CD8 TEMRa HLA-DR percentage, therefore the number of participants analyzed was reduced from 25 to 23 participants.
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRa HLA-DR T cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRa HLA-DR T cells | 3.69 (2.97)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Baseline and Week 48; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 3.69, 95% CI 2-sided [2.40 to 4.97], Standard Deviation 2.97 — Difference was calculated as Baseline minus Week 48

52. Secondary Outcome: Difference in CD8 TEMRa HLA-DR Percentage Between Week 48 and Week 152
Time Frame: 152 weeks
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: percentage of CD8 TEMRa HLA-DR T cells
Arm/Group | Experimental Arm
Number analyzed (Participants) | 23
percentage of CD8 TEMRa HLA-DR T cells | -1.31 (2.54)
Statistical Analysis 1: Comparison: Experimental Arm; Null hypothesis is no changes between Week 48 and Week 152; Test type: Superiority or Other; p = 0.0215, t-test, 2 sided; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-2.41 to -0.21], Standard Deviation 2.54 — Difference was calculated as Week 48 minus Week 152

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 152 week period.
Description: Subjects were assessed for adverse events at each study visit.
Arm/Group | Experimental Arm | Standard Care Arm
Serious Adverse Events (participants affected / at risk) | 2/75 | 1/27
Other Adverse Events (participants affected / at risk) | 9/75 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=75) | Standard Care Arm (N=27)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutriphil Count Decreased (Investigations) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=75) | Standard Care Arm (N=27)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 0 (0)
Blood Bilirubin Increased (Investigations) | 4 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.